CLINICAL TRIAL: NCT03395626
Title: Validity and Safety of Symptom Improvement of ID-JPL934 for Abnormal Bowel Movement Such as Constipation, Diarrhea, Abdominal Pain: Randomized, Double-blind, Placebo-controlled, Parallel-group Study
Brief Title: ID-JPL934 for Abnormal Bowel Movement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ID-JPL934
Record Dates: First submitted 2018-01-04; First posted 2018-01-10 (Actual); Last update posted 2018-01-30 (Actual); Status verified 2017-08

CONDITIONS: Abnormal Bowel Movement Such as Constipation, Diarrhea, Abdominal Pain
MeSH Terms: conditions — Diarrhea; Abdominal Pain

STUDY DESIGN:
Intervention Model Description: randomized, double-blind, placebo-controlled, parallel-group
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ID-JPL934 (Experimental): probiotics 20%, corn starch 80%
  Interventions: Dietary Supplement: ID-JPL934
- placebo (Placebo Comparator): corn starch 100%
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: ID-JPL934 — probiotics
  Arms: ID-JPL934
Dietary Supplement: Placebo — corn starch
  Arms: placebo

SUMMARY:
Probiotics, which are part of the human body, are microorganisms, which are known to have beneficial effects when consumed in a certain amount, and have the function of controlling intestinal flora and inhibiting inflammation. Recently, probiotics have received much attention in the treatment of hypersensitivity syndrome. The aim of this study was to investigate the effect of probiotic strains, ID-JPL934, in the diagnosis of irritable bowel syndrome.

Overall satisfaction with improvement of bowel habits such as diarrhea and constipation as well as abdominal discomfort and abdominal discomfort in the group receiving ID-JPL934 capsules (test food group or test group) and control group (control food group or control group) (0-10 point visual analogue scale) for each symptom before and after ingestion to evaluate the degree of improvement of the symptoms. The purpose of this study was to investigate the relationship between bacterial composition changes in the stool and the improvement of symptoms in the patients before and after ingestion.

ELIGIBILITY:
Inclusion Criteria:

1. Korean men and women aged over 19 and 80
2. Adults with the following criteria (1) If the symptoms are relieved by bowel movements and changes in the number of bowel movements with less than two stomach complaints or stomach complaints every three months (2), these two forms of bowel movements have started (3)
3. Methodological-fractive women or fertile women who are negative during pregnancy diagnostic tests (urine or seron- hCG). An appropriate method of birth control (e.g., " oral contraceptive " or bi-fertility) during an examination
4. People who have no problems in their nerves and mental systems and who can make their own doctors clear
5. The person who agreed in writing to this test

Exclusion Criteria:

1. Persons with hypersensitivity to probiotics
2. Pregnant or lactating women
3. People who have received other clinical trial drugs within the first 3 months of visit 1. However, in the case of lactic acid bacteria preparation, the test can be taken after a two week absence period.
4. A person who believes that the participant is in a condition or situation in which participation in the clinical trial may be hazardous to the participant,
5. Patients with severe congestive heart failure or severe angina
6. If the patient is diagnosed as having urticaria or immunosuppression
7. Patients who are taking or taking medications (formulants, lactic acid bacteria) that may affect the test food, probiotics, or during the test period. However, if you are taking the drug, you can take the test after two weeks of abstinence.
8. If the systolic blood pressure measured at Visit 1 is greater than 160 mmHg or diastolic blood pressure is greater than 100 mmHg and hypertension is not controlled regardless of whether the medication is administered or not.
9. Patients with uncontrolled endocrine diseases (such as diabetes), metabolic diseases (eg secondary hyperlipidemia) or hypothyroidism (subjects with a history of hypothyroidism) should receive a stable thyroid hormone supplement for at least 4 weeks prior to visit 1 If you are on therapy, you can participate in this test only if the TSH level measured at Visit 2 is within the normal range.)
10. If kidney function is impaired at visit 1 (creatinine> 2.0 mg / dL) or nephrotic syndrome is observed
11. If the cancer has developed within the past 5 years (unless it is determined to be cured)
12. If there is a history of mental instability and drug / alcohol abuse within the past 5 years, or if major psychiatric illnesses are not adequately controlled and stabilized by medication
13. Visits 1 If you have taken mental nerve agents within the previous 3 months
14. If you take a systemic steroid preparation within 1 month before visit 1
15. Patients who underwent abdominal surgery except for appendectomy, hernia surgery, and cesarean section
16. People who are suffering from hypersensitivity syndrome in the ROME Ⅲ standard
17. Any person deemed inappropriate for the judgment of the clinician

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2017-07-12 (Actual); Primary Completion 2017-10-02 (Actual); Study Completion 2018-03-31 (Estimated)

PRIMARY OUTCOMES:
symptom improvement effect | 8week
  symptom questionnaire survey

SECONDARY OUTCOMES:
VAS score | 8week
  Visual analogue scale score(10-point scales)
QoL score | 8week
  Quality of Life score (5-point scales)

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bungdang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shin CM, Choi YJ, Lee DH, Moon JS, Kim TY, Kim YK, Lee WH, Yoon H, Park YS, Kim N. Validity and safety of ID-JPL934 in lower gastrointestinal symptom improvement. Sci Rep. 2021 Jun 22;11(1):13046. doi: 10.1038/s41598-021-92007-3. PMID 34158518